## **NORTH STUDY:**

A Phase II Study of Panobinostat in Paediatric, Adolescent and Young Adult Patients with Solid Tumours Including Osteosarcoma, Malignant Rhabdoid Tumour/Atypical Teratoid Rhabdoid Tumours and Neuroblastoma

# **Statistical Analysis Plan**

V1.0 December2024

Protocol: ACCT008/ASSG35
ClinicalTrials.gov ID: NCT04897880
Novartis Ref: CLBH589XAU13T
Based on protocol Version 5, dated 18Sept2020

#### Alannah Rudkin.

Clinical Epidemiology & Biostatistics Murdoch Children's Research Institute The Royal Children's Hospital, 50 Flemington Road Parkville, Victoria 3052 Australia

**CONTENTS** 

**Table of Contents** 

| 1. Administrative Information | 3 |
|------------------------------------|----|
| 1.1 Document Version History | 3 |
| 1.2 Approvals | 4 |
| 2. Study Synopsis | 4 |
| 2.1 Objectives | |
| 2.1.1 Primary Objectives | 6 |
| 2.1.2 Secondary Objectives | 6 |
| 2.2 Endpoints | 6 |
| 2.3 Study Population | 7 |
| 2.4 Intervention | 8 |
| 2.5 Randomisation And Blinding | 9 |
| 2.6 Sample Size | 9 |
| 2.7 Study Procedures | 9 |
| 3. General Statistical Methodology | 11 |
| 3.1. Scope | |
| 3.2. Analysis Software | |
| 3.3. Data Verification | |
| 3.4. Definition Of Baseline | |
| 3.5. Assessment Of Response | |
| 3.6. Adverse Events | |
| 3.7. Year, Month And Duration | |
| 4. Descriptive Statistics | |
| 4.1. Recruitment And Follow-Up | |
| 4.2. Baseline Characteristics | |
| 4.3. Protocol Deviations | |
| 4.4. Compliance | |
| 4.5. Concomitant Therapies | |
| 5.1. Main Analysis | |
| 5.1.1 Event Free Survival | |
| 5.1.2. Overall Survival | |
| 5.1.3 -Safety | |
| 6. Secondary Endpoints | |
| 6.1 Main Analysis | |
| 6.1.1 Clinical Benefit Rate | 19 |
| 7. Exploratory Outcomes | 21 |
| 7.1 Comparison To Historical Data | 21 |
| 8. Missing Data | |
| 9. Listings, Tables And Figures | |
| 9.1. List Of Listings | |
| 9.2. List Of Tables | |
| 9.3. List Of Figures | 22 |

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

AE Adverse Event

ATRT Atypical Teratoid Rhabdoid Tumour

CBR Clinical Benefit Rate
CR Complete Response
Cl Confidence Interval
CNS Central Nervous System

CRF Case Report Form

CT Computed tomography scan

DLT Dose Limiting Toxicity

DSMC Data Safety Monitoring Committee

FDG-PET fluorodeoxyglucose positron emission tomography

GCP Good Clinical Practice

INRC International Neuroblastoma Response Criteria

ITT Intent-To-Treat

MRT Malignant Rhabdoid Tumour MRI

Magnetic resonance imaging
OS Overall survival
PR Partial Response

PMNC Peripheral Mononuclear Cells

PD Progressive Disease

RT Radiotherapy

RANO Response Assessment in Neuro-Oncology
RECIST Response Evaluation Criteria in Solid Tumours

SAE Serious Adverse Event
SD Standard Deviation
SE Standard Error

SSI Significant Safety Issue

SD Stable Disease

SUSAR Suspected Unexpected Serious Adverse Reaction

TTP Time to progression

## 1. ADMINISTRATIVE INFORMATION

Protocol: ACCT008/ASSG35; Version 5; 18Sep2020

Novartis Ref: CLBH589XAU13T

ClinicalTrials.gov Identifier: NCT04897880

## 1.1 Document Version History

| Version Date | Version | Author | Signature | Change Description | Reason/Comment |
|---|---|---|---|---|---|
| December<br>2024 | 1.0 | AR | pour | Initial release. | Not applicable. |

Protocol: ACCT008/ASSG35

#### 1.2 Approvals

The undersigned have reviewed this plan and approve it as final. They find it to be consistent with the requirements of the protocol as it applies to their respective areas. They also find it to be compliant with ICH-E9 principles and confirm that this analysis plan was developed in a completely blinded manner (i.e. without knowledge of the effect of the intervention being assessed)

| Name | Role on Study | Affiliation | Signature | Date |
|---|---|---|---|---|
| Prof David Ashley | Study Chair | The Preston Robert Tisch Brain Tumor Centre Duke University Medical Centre | al- | 21Aug2024<br>(draft reviewed,<br>unable to review<br>December 2024<br>version) |
| A/Prof Jayesh | Study Chair | Drug Development Group | | |
| Desai | | Peter MacCallum Cancer Centre | Ayinthayesir Desemblan 6,2025 (6,46 Gillin 211) | 06/01/25 |
| Dr Paul Wood | Study Chair | Children's Cancer Centre, Monash<br>Children's Hospital, Monash<br>Health | (Mun) | 16Dec2024 |
| Alannah Rudkin | Statistician | Murdoch Children's Research<br>Institute | prolin | 09Dec2024 |

#### 2. STUDY SYNOPSIS

This is a multi-centre, open-label, single-arm Phase 2 study in participants < 40 years old with refractory solid and CNS tumours. Participants were stratified by tumour type: osteosarcoma, neuroblastoma, and malignant rhabdoid tumour or atypical teratoid rhabdoid tumours (ATRT/MRT). Eligible participants included those with refractory or relapsed osteosarcoma, neuroblastoma and MRT/ATRT, or newly diagnosed MRT/ATRT that were stable after completion of standard therapy. Participants must have had histologic verification of the diagnosis of malignancy at either the time of initial diagnosis or at relapse. A maximum of 60 participants (20 per strata) were planned to be treated with panobinostat as a continuous oral dose starting at 10 mg/m² per day. Study treatment was planned to continue until disease progression, intolerable toxicity, or participant decision for a maximum of one year (12 treatment courses of 28 days duration each). Patients will be followed for up to 2 years from completion of study therapy.

The study design schematic is presented in Figure 2.1-1



#### **Schedule of Analyses:**

The dose evaluation and study expansion analyses in each strata were evaluated separately to this SAP. They are described below.

#### **Dose Evaluation**

The biological activity of panobinostat at a given dose level was determined by the real-time acetylation status (as defined by acetylated H4 on Peripheral Mononuclear Cells (PMNC)s) at day eight compared with pre-treatment. This analysis was performed for a minimum of 2 patients in each strata at the required dose levels. Once biological activity was confirmed via the acetylation status of H4 on PMNC at any dosing level in any strata, it did not need to be repeated and dosing adjustments could be made on dose limiting toxicities (DLTs) and adverse events (AEs) alone.

i) If significant increase in acetylation, and therefore biological activity, was demonstrated at the starting dose of 10 mg/m² then no dosing adjustment took place unless DLTs/AEs were observed. ii) In the case of drug toxicity and irrespective of biological activity, intra-patient dose reductions in 2 mg/m² increments were applied, and the dose level for the strata reviewed. iii) In the case of inadequate biological activity, with no toxicity, intra-patient dose escalations of 2 mg/m² were recommended.

The final dose per strata was the level where continuous dosing was maintained for a 4-week period with acceptable toxicity and biological effect. The final Panobinostat doses were 6mg/m2 per day for the ATRT/MRT cohort, 8mg/m2 per day for the neuroblastoma cohort, and 4mg/m2 per day for the osteosarcoma cohort.

## Study Expansion

Protocol: ACCT008/ASSG35

The study employed a Simon two-stage minimax design (1). At trial design stage an initial efficacy analysis was planned when a minimum of 9 patients in each strata were enrolled. The regimen would be considered worthy of further study if disease stability at 4 months was observed in 3 or more of the first 9 patients in a stratum and less than 30% of patients experience a DLT at the final dose level. If this was achieved, recruitment would proceed to a total of 20 patients in each strata.

However, due to uncertainty of panobinostat supply, a decision was made to permanently close the osteosarcoma and neuroblastoma arms prior to the initial efficacy analysis when 9 and 2 had been enrolled in the osteosarcoma and neuroblastoma arms, respectively. At that time, it was decided to continue recruitment into the ATRT/MRT cohort who had met the initial efficacy criteria for 3/9 participants with disease stability and <30% experiencing a DLT at the final dose level. The ATRT/MRT arm closed in December 2021 due to termination of the study supply agreement, at that time 14 participants had been enrolled in the ATRT/MRT arm.

#### 2.1 OBJECTIVES

#### 2.1.1 PRIMARY OBJECTIVES

The primary aims of this study are as follows:

- a) To define the anti-tumour activity of low dose continuous panobinostat.
- b) To define and describe the toxicities of panobinostat for patients on a continuous dosing schedule.

#### 2.1.2 SECONDARY OBJECTIVES

The secondary aims are:

- a) To define the anti-tumour activity of low dose continuous panobinostat using functional imaging techniques.
- b) To assess the biologic activity of low dose panobinostat by measuring histone acetylation status in peripheral mononuclear cells (PMNC), bone marrow and fresh tumour tissue specimens in all patients (when available).

#### 2.2 ENDPOINTS

#### 2.2.1 PRIMARY ENDPOINTS

- a) Estimated 2-year Event free survival (EFS). EFS is calculated as the time from study enrolment to first documented disease progression, relapse or second malignancy, or death from any cause
- b) Estimated 2-year Overall Survival (OS). OS is calculated as the time from study enrolment to death from any cause.
- c) Safety, as assessed by incidence of adverse events graded according to the NCI-CTCAE, version 4.0 [Time Frame: 1 week to 12 months after intervention commencement]

#### 2.2.2 SECONDARY ENDPOINTS

a) Efficacy as measured by Clinical Benefit Rate (percentage of patients with stable disease or better using MRI/CT imaging) at 6 and 12 months after intervention commencement. Stable disease is defined as MRT/ATRT/Osteosarcoma with complete response (CR), partial response (PR), minor response (MR), stable disease (SD) overall response. Neuroblastoma with CR/PR/SD or Non-CR/Non-PD overall response.

#### 2.2.3 EXPLORATORY ENDPOINTS

a) Comparing overall and event free survival for ATRT patients to historical data. Comparison of EFS and OS up to 2 years post enrolment.

#### 2.3 STUDY POPULATION

#### Inclusion criteria:

- Patients must be < 40 years of age.</li>
- Patients with refractory or relapsed osteosarcoma, neuroblastoma and MRT/ATRT or newly diagnosed MRT/ATRT. Patients must have had histological verification of the diagnosis of malignancy at time of diagnosis or relapse.
- Patient's disease is considered refractory, according to their treating hospital standard practice guidelines, to conventional therapy except for newly diagnosed ATRT/MRT. This includes relapsed patients who may be off treatment. Patients must have stable disease (SD) or better.
- Karnofsky ≥ 60% for patients ≥ 16 years of age, <u>OR</u> Lansky ≥ 60% for patients < 16 years of age.</li>
- Life expectancy of greater than 8 weeks.
- Fully recovered from acute toxic effects of all prior chemotherapy, immunotherapy or radiotherapy prior to entering study.
- Patients with CNS tumours who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week.
- Adequate BM function peripheral ANC  $\geq$  750/µl (0.75 x 10<sup>9</sup>/L); platelet count  $\geq$  75,000/µl (75 x 10<sup>9</sup>/L); haemoglobin  $\geq$  8g/dL (80 g/L).
- Adequate renal function age-adjusted normal serum creatinine or GFR > 70ml/min/1.73m<sup>2</sup>.
- Adequate liver function total bilirubin  $\leq 1.5 \times IULN$  for age, ALT  $\leq 5 \times IULN$  for age, and albumin  $\geq 2g/dL$  (20g/L).
- Adequate cardiac function shortening fraction of ≥ 27% OR ejection fraction of ≥ 50% by echocardiogram.
- Adequate respiratory function defined as no evidence of dyspnoea at rest, no exercise intolerance and pulse oximetry (SaO<sub>2</sub>) > 94% in room air.
- Adequate CNS function seizure free for 2 months.

- Adequate serum calcium, magnesium, and potassium concentrations all must be ≥ ILLN for age, with or without supplementation.
- If female and post-menarcheal, pregnancy test must be negative.
- If of reproductive potential, have agreed to use effective contraceptive method.
- If female and lactating, have agreed not to breastfeed.
- Patient and/or their legal representative have signed a written informed consent form.

#### Exclusion criteria:

- Patients who have received myelosuppressive chemotherapy and/or biologic therapy within 3 weeks (4 weeks if prior nitrosourea).
- Patient has received local palliative radiotherapy within 2 weeks.
- Patient has received craniospinal radiotherapy within 3 weeks.
- Patient has received ≥ 50% radiation of pelvis within 6 weeks.
- Patient has received other substantial BM radiation within 6 weeks.
- Have received growth factor(s) within 1 week.
- Are receiving enzyme inducing anticonvulsant therapy. In order to be eligible, patients
  must be transferred to and stabilised on an eligible anticonvulsant as listed in Appendix II
  as per local institutional practice. (See Appendix II for a list of enzyme inducing and
  nonenzyme inducing anticonvulsants).
- Are on medications associated with prolongation of QTc interval as listed in Appendix III.
- Are receiving hydrochlorothiazide.
- Are receiving metronidazole and/or disulfiram. This is due to the increased risk of metabolic acidosis when patients are concomitantly on panobinostat and metronidazole and/or disulfiram.
- · Patients with uncontrolled sepsis.
- Patients who have previously received panobinostat.
- Patients with symptoms of congestive heart failure, uncontrolled cardiac rhythm disturbance, or a QTc (Fridericia's formula) that is > 450 msec.

#### 2.4 INTERVENTION

A three-week washout period was required after conventional myelosuppressive chemotherapy and/or biologic therapy to start Panobinostat therapy.

Panobinostat was supplied in capsule form and administered orally. Each course consisted of 4 weeks (28 days). Treatment will continue for up to 12 months consisting of 12 treatment courses, each of 4 weeks (28 days) duration.

Intra-patient dose adjustments of 2 mg/m<sup>2</sup> were made to a starting dose of 10 mg/m<sup>2</sup> based on DLTs/AEs and biological activity, and dose level for that stratum reviewed. For full criteria for dose escalation and reduction see protocol version 5.0 18Sep2020. The final dose per strata was the level where continuous dosing is maintained for a 4-week period with acceptable toxicity and biological effect.

Protocol therapy could be terminated for the following reasons: a) Progressive disease (radiographic or clinical)

b) Irreversible or unacceptable dose-limiting toxicity

c) Other adverse event

Protocol: ACCT008/ASSG35

- d) Refusal of further protocol therapy by patient or parent/guardian
- e) Physician determines it is not in the patient's best interest
- f) Pregnancy
- g) Termination or suspension of clinical trial

The investigator's clinical judgment was used to determine whether a subject should be removed from treatment or from the study due to progressive disease, AE or DLT, or another reason.

#### 2.5 RANDOMISATION AND BLINDING

This a single arm open label study.

#### 2.6 SAMPLE SIZE

The study employed a Simon two-stage minimax design (1). A 30% gain in Clinical Benefit Rate (CBR) was considered as the minimum gain required to warrant further study of this regimen. In this case the clinical benefit to be observed is stability of disease. 70% stability at 4 months would be indicative of clinical utility, whereas a rate of 40% would be the lower limit of interest, with  $\alpha$  = .15 and  $\beta$  = .10. The minimal accrual number required in each strata was 14 patients. This was increased to 20 patients in each strata, over 3 years, for a total of 60 patients.

The biological activity analysis was performed for a minimum of 2 patients in each strata at the required dose levels.

#### **2.7 STUDY PROCEDURES**

All entry requirements had to be completed during the four-week screening period before study enrolment.

| Studies to be Obtained | Pre-salvage<br>therapy <sup>a</sup> | Screening<br>prior to<br>enrolment<br>(Baseline) | Weeks 1-4<br>(first 28 day<br>course) | Subsequent<br>Months<br>(28 day courses) | Follow-up <sup>b</sup> |
|---|---|---|---|---|---|
| History (including AEs/DLTs) | | Х | Weekly | Х | Х |
| Physical Exam (height, weight, BSA) | | х | Weekly | х | х |
| Performance Status<br>Refer to Appendix I | | Х | Weekly | х | х |
| Full Blood Evaluation (FBE) with Differential & Blood Film | | Х | Weekly | Х | х |
| Urinalysis <sup>c</sup> | | Х | Weekly | х | |
| Urea & Electrolytes<br>Calcium, Magnesium & Potassium | | Х | Weekly | х | х |
| Renal Function/GFR/Creatinine | | Х | Weekly | Х | х |
| Liver Function Tests including Total Protein & Serum Albumin | | х | Weekly | х | Х |

| Thyroid Function Tests (TFTs including TSH, T3, T4) | | X | | End of therapy | |
|---|---|---|---|---|---|
| CT/MRI of Primary Tumour <sup>d</sup> | х | х | | 2 monthly | X e |
| MRI Spine (ATRT only) Refer to Section | Х | х | | 2 monthly <sup>f</sup> | X e,f |
| FDG-PET/DOTATATE 8 | х | х | | 2 monthly | X e |
| MIBG<br>(Neuroblastoma only) | х | х | | 2 monthly | X e |
| CXR<br>(ATRT only) | Х | X h | | End of therapy | |
| Abdominal Ultrasound<br>(ATRT only) | Х | X h | | End of therapy | |
| MRI Brain<br>(MRT only, not primary site) | Х | X h | | End of therapy | |
| CT Chest / CXR<br>(Osteosarcoma only, non-lung primary) | Х | X (CT and<br>CXR) | | 2 monthly<br>(CXR, CT and CXR<br>at end of therapy) | X<br>(CT or CXR) |
| Blood Samples – HDACi<br>[Not applicable to United States] | | Pretreatment | 7 days after first<br>dose | | |
| Bone Marrow Evaluation (only if clinically indicated) including HDACi studies [Not applicable to United States] | | Х | End of Course | If positive at<br>baseline or as<br>clinically indicated | |
| Pregnancy Test <sup>i</sup> | | х | | | |
| ECG | | Х | End of Course | Х | |
| Echocardiogram | | Х | | 6 monthly | |

- a If applicable and where available, these will be the last set of imaging investigations performed as part of routine patient care prior to salvage therapy.
- b Up to 2 years from completion of therapy. c Not mandated at every time point, urinalysis performed per institutional practice.
- d Use the same imaging modality throughout the course of the study e Follow-up imaging studies are not required if there is documented evidence of overt clinical progression. Follow-up imaging is 3 monthly or per routine follow-up.
- f Repeat Spine MRI only if initially positive
- g Use FDG-PET in non-CNS MRT.

Protocol: ACCT008/ASSG35

- Use FDG-PET in all osteosarcoma and neuroblastoma (if not MIGB avid).
- Could be DOTATATE scans in neuroblastoma patients, when available, following discussion with Study Chair.
- h Scans performed outside the four-week screening period as standard of care, are acceptable.
- i Females of child-bearing age required a negative pregnancy test prior to entering study.

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

j Follow-up for participants remaining on study was every 6 weeks for the first 3 months, then every 3 months for up to 2 years from completion of therapy. Patients may needed to be seen more frequently than these defined intervals based on their medical needs.

In instances where participants discontinued study drug before completion of therapy, they were encouraged to continue with study follow-up visits as long as such procedures did not pose a risk to the well-being of the patient.

#### Measurement of effect

#### Survival Measure

At each study visit (every 28 days) while on treatment, patient study status will be collected. If a patient terminates treatment early, the reason and date will be collected. This includes progressive disease, toxicity or adverse event, and death.

Follow-up for participants remaining on study will be every 6 weeks for the first 3 months, then every 3 months for up to 2 years from completion of therapy.

After treatment completion, patient death or lost to follow up will be collected at follow up visits.

#### **Event Measure**

Radiographic progressive disease will be captured in the overall response at each disease assessment as per section 9 of protocol. Clinical progression will be documented during study visits as described above.

Full details of the background to the trial and its design are presented in the protocol.

### 3. GENERAL STATISTICAL METHODOLOGY

#### 3.1. SCOPE

The biological activity analysis was performed during the trial to determine dosing levels (real time acetylation data). This analysis and its results are not in the scope of this analysis. See section 4.3 of protocol for more information.

#### 3.2. ANALYSIS SOFTWARE

All analyses will be performed using Stata Release 18 or later.

#### 3.3. DATA VERIFICATION

All variables included in analysis will be assessed for validity. Range checks will be performed on all continuous variables. Categorical variables will be assessed for consistency with the protocol and relevant data dictionary. Any data verification queries will be raised with the study team.

#### 3.4. DEFINITION OF BASELINE

Baseline will be defined period between consent date and date of enrolment.

NORTH: Statistical Analysis Plan 

Date of enrolment (day 0) will be the eligibility visit date in the database, visdat.

Baseline values used to define changes in measurements over time for each participant are defined as the closest to and including day 0 within the preceding 28 days. Where more than one measurement is available within this window the closest to enrolment will be used.

Patients were enrolled on the study once all eligibility requirements for the study were met. The National Coordinating Centre, in conjunction with the Study Chair, reviewed the submitted eligibility information and supporting source documentation.

Start of treatment is defined as (Week 1 Day 1 visdat) from the study status database.

#### 3.5. ASSESSMENT OF RESPONSE

Protocol: ACCT008/ASSG35

The revised Response Evaluation Criteria in Solid Tumours (RECIST), Version 1.1, will be used to evaluate tumour response for non-CNS solid tumours. The Response Assessment in NeuroOncology Working Group's updated response assessment criteria (RANO) will be used to evaluate tumour response for CNS solid tumours. The revised International Neuroblastoma Response Criteria will be used to evaluate tumour response for neuroblastoma. For further details of these definitions please refer to the protocol.

The study investigator's evaluation of overall response will be used in analysis.

#### 3.6. ADVERSE EVENTS

Adverse events will be coded according to the Common Terminology Criteria for Adverse Events V4.0 (CTCAE V4.0).

#### 3.7. YEAR, MONTH AND DURATION

The following conversion factors will be used to convert days to months or years: 1 month =30.4375 days, 1 year = 365.25 days. Duration will be calculated as (end date – start date + 1).

#### 4. DESCRIPTIVE STATISTICS

Analysis will be completed by disease strata;

MRT/ATRT (strata 1), osteosarcoma (strata 2), or neuroblastoma (strata 3).

#### 4.1. RECRUITMENT AND FOLLOW-UP

A CONSORT flowchart of patient enrolment and follow up will be provided.

The number of patients and the proportions who were consented, screen failed, enrolled, completed treatment, and completed follow-up will be summarised by disease strata.

#### 4.2. BASELINE CHARACTERISTICS

Patient and disease characteristics at baseline will be summarised by disease strata. Continuous variables will be reported with mean with range and categorical variables will be reported with frequencies and proportions. For neuroblastoma, results for the two individual patients will be reported. A listing of all characteristics for each patient will be provided.

This will include number with study indication (MRT/ATRT, osteosarcoma, neuroblastoma), disease event (newly diagnosed, relapsed, refractory, un-resectable lesion), number of relapse if applicable, disease status (stable disease, remission), central nervous system (CNS) disease, best response to prior treatment, prior surgery, prior chemotherapy, prior radiotherapy (RT) and location, RT total dose (Gy) if applicable, and other prior treatment.

Patient demographics summarised will include age, sex, ethnicity, indigenous status, and baseline performance score (Karnofsky  $\geq$  16 years old, Lansky < 16 years old).

#### 4.3. PROTOCOL DEVIATIONS

Protocol deviations will be listed and summarised by disease strata.

#### 4.4. COMPLIANCE

Mean (range) number of treatment courses completed (28 days per cycle) and time in follow up (weeks) will be summarised by disease strata. The number of patients who completed each course (full 28 days) will be listed for each disease strata, with reasons for early treatment termination listed.

Panobinostat dose (mg/m²) days compliant, and total days of treatment will be summarised by mean and range by disease strata. A summary of dose received by treatment course will also be listed.

#### 4.5. CONCOMITANT THERAPIES

All medications and significant non-drug therapies will be recorded throughout the study period. This includes medications commenced from 14 days before until 28 days after the study drug is administered. Medications include both prescribed and over the counter (OTC) medications including herbal and vitamin treatments.

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

A listing of concomitant medications will include medication name and reason sorted by disease strata.

#### 5. ANALYSIS OF THE PRIMARY OUTCOME(S)

#### 5.1. MAIN ANALYSIS

#### 5.1.1. Event free survival

## **Primary Estimand**

**Population**: All patients eligible and enrolled into trial with MRT/ATRT (strata 1), osteosarcoma (strata 2), or neuroblastoma (strata 3).

**Treatment**: Panobinostat

**Outcome**: Estimated 2-year Event free survival (EFS). EFS is calculated as the time from study enrolment to first documented disease progression, relapse or second malignancy, or death from any cause up to 2 years after study enrolment. The latest possible time of risk being 2 years after enrolment, or the last date known alive.

**Summary measure**: The probability of EFS (Kaplan-Meier) at with 95%CI will be estimated each stratum\*. Kaplan- Meier curves will be plotted for EFS probability, enrolment date as start of risk period. Median EFS time will be calculated at 2 years post-enrolment.

#### **Subgroup Analysis:**

Descriptive statistics (proportions) by subgroup for each disease strata.

Age at enrolment <36 months (3 years old) vs. ≥36 months Radiation therapy (RT) vs. no RT Disease status at trial entry (complete response vs stable disease)

#### **Intercurrent Events**

#### **Potential intercurrent events:**

Patient comes off study or treatment due to toxicity before an event is observed. Patient comes off study or treatment to receive another treatment.

#### Strategy for handling intercurrent event:

#### **Treatment policy**

EFS will be estimated for patients regardless of early treatment or trial termination. This approach assumes that data collected is reflective of those missing data (patients who withdrew from trial).

#### **Sensitivity Analysis**

#### **Composite Strategy**

Patients coming off study or protocol treatment due to an irreversible or unacceptable dose limiting toxicity or a Serious adverse event (SAE) before an event is observed, will be handled by the composite strategy. The removal from study/treatment date will be treated as an event.

only calculated if stratum had adequate sample size (osteosarcoma and ATRT/MRT only).

Protocol: ACCT008/ASSG35

Patients coming off study or protocol treatment to receive another treatment will also be handled by this strategy in the same analysis.

#### **Primary Estimand Calculation**

EFS will be estimated and visualised using the Stata sts list and graph commands.

stset tvar, fail(event) origin(time enrol\_date) enter(time consent\_date) sts list, strata(disease type) risk table(6 12 24) sts graph, strata(disease type) risk table(0 6 12 18 24) xlabel(0 6 12 18 24) tmax(24) Median EFS will be estimated using Stata stsum command stsum, by(disease type)

#### Subgroup analysis

The proportion in each group and 95%CI will be estimated using Statas ci proportions command.

Sensitivity analysis ( as above with alternate event) *stset tvar,* fail(event\_comp) origin(time enrol\_date) enter(time consent\_date)

Where time is in months and patients will be censored at their last known contact alive.

#### 5.1.2. Overall survival

#### **Primary Estimand**

**Population**: All patients eligible and enrolled into trial with MRT/ATRT (strata 1), osteosarcoma (strata 2), or neuroblastoma (strata 3).

**Treatment**: Panobinostat, dosing as per protocol.

**Outcome**: Estimated Overall Survival (OS). OS is calculated as the time from study enrolment to death from any cause.

**Summary measure**: The OS probability (Kaplan-Meier) and 95%CI will be estimated for each stratum\* up to 2 years post- enrolment. Kaplan- Meier curves will be plotted for OS probability; enrolment date as start of risk period. The number of deaths and the median OS time will be reported up to 2 years post-enrolment.

#### **Subgroup Analysis:**

As per section 5.1.1

#### **Intercurrent Events**

#### **Potential intercurrent events:**

Patient comes off study due to toxicity, or to start a new treatment.

#### Strategy for handling intercurrent event:

<sup>\*</sup>only calculated if stratum had adequate sample size (osteosarcoma and ATRT/MRT only).

Protocol: ACCT008/ASSG35

Patients coming off study due to a related toxicity or to start a new treatment will be handled with the treatment policy. OS will be analysed for all patients regardless of treatment received until last study visit.

#### **Sensitivity Analysis**

#### **Composite Strategy**

Patients coming off study due to toxicity or to start a new treatment before death could be observed will be handled by the composite strategy. The removal from study date will be treated as an event/death in sensitivity analysis.

#### **Estimand Calculation**

OS will be estimated and visualised using the Stata sts list and graph commands. stset tvar, fail(death) origin(time enrol\_date) enter(time consent\_date) sts list, strata(disease type) sts graph, strata(disease type) tmax(24) Median OS will be estimated using Stata stsum command stsum, by(disease type)

Where time is in months and patients will be censored at their last known contact alive.

#### 5.1.3 -Safety

Adverse events will be summarised by grade and type defined by CTCAE Version 4 from 1 week to 12 months after intervention commencement.

Relationship to study drug (definite, probable, possible) adverse events summarised in a table, with the worst AE grade reported by each participant.

A summary table of Dose Limiting Toxicities will include AE type, grade, and frequency.

#### 6. SECONDARY ENDPOINTS

Protocol: ACCT008/ASSG35

## Measurement of effect

Evaluation of disease will be conducted by the investigator as outlined in the protocol. Stable disease will be confirmed on study entry, and tumour response determined at each imaging assessment time point. Overall response as determined by the investigator will be used for the secondary efficacy outcome analysis.

<u>Response Assessment for Non-CNS Solid Tumours</u> - Osteosarcoma and MRT The revised Response Evaluation Criteria in Solid Tumours (RECIST), Version 1.1, will be used to evaluate tumour response, as assessed by medical imaging.

#### Overall Response for Non-CNS Tumours (Measurable Disease)

| . Target lesions | Non-target lesions | New lesions | Overall response |
|------------------|--------------------|-------------|------------------|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| | Non-CR/non-PD/ | | |
| PR | Not evaluated | No | PR |
| S.D. | Non-CR/non-PD/ | | <b>an</b> |
| SD | Not evaluated | No SD | SD |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |
| Not evaluated | Non-PD | No | Inevaluable |

Overall Response for Non-CNS Tumours (Non-Measurable Disease)
Non-target New Overall lesions lesions
response

| CR | No | CR |
|-------------------|--------------|------------------|
| Non-<br>CR/non-PD | No | Non-<br>CR/nonPD |
| Not all evaluated | No | Inevaluable |
| Unequivocal<br>PD | Yes or<br>No | PD |
| Any | Yes | PD |

## Response Assessment for CNS Solid Tumours- ATRT

The Response Assessment in Neuro-Oncology Working Group's (RANO) updated response assessment criteria, will be used to evaluate tumour response. Overall response will be defined by the response of the individual components – contrast enhancing lesions, non-enhancing lesions, new lesions, corticosteroids, and clinical status per the investigator at each imaging timepoint.

| Complete | Requires <u>all</u> the following | criteria to be met: |
|---|---|---|
| Response<br>(CR) | Contrast enhancing disease | Complete Response: Complete disappearance of all measurable and non-measurable disease |
| | New lesions | No new lesions |
| | Non-enhancing lesions | Stable or improved T2/FLAIR lesions |
| | Corticosteroids | Patient off corticosteroids (or on physiologic replacement doses only) |
| | Clinical Status | Stable or improved clinically |
| Partial | Requires all the following | |
| Response<br>(PR) | Contrast enhancing disease | Partial Response: ≥ 50% decrease, compared with baseline, in the sum of products of perpendicular diameters of all measurable enhancing lesions |
| | Name In all and | No progression of non-measurable disease No new lesions |
| | New lesions Non-enhancing lesions | Stable or improved T2/FLAIR lesions on the same or lower dose of corticosteroids compared with baseline scan |
| | Corticosteroids | Corticosteroid dose at the time of evaluation no greater than the dose at time of baseline scan |
| | Clinical Status | Stable or improved clinically |
| Stable | Requires <u>all</u> the following | criteria to be met: |
| Disease (SD) | Contrast enhancing disease | Stable Disease: Does not qualify for complete response, partial response, or progression |
| | New lesions | No new lesions |
| | Non-enhancing lesions | Stable T2/FLAIR lesions on the same or lower dose of corticosteroids compared with baseline scan |
| | Corticosteroids | Corticosteroid dose at the time of evaluation no greater than the dose at time of baseline scan |
| | Clinical Status | Stable or improved clinically |
| Progressive | Defined by <u>any</u> of the foll | owing: |
| Disease (PD) | Contrast enhancing disease | Progressive Disease: ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumour measurement obtained at baseline (if no decrease) or best response, on stable or increases doses of corticosteroids Clear progression of non-measurable disease |
| | New lesions | Any new lesion |
| | Non-enhancing lesions | Significant increase in T2/FLAIR lesions on stable or increasing doses of corticosteroids, not caused by comorbid events |
| | Corticosteroids | N/A * |
| | Clinical Status | Clear clinical deterioration not attributable to other causes apart from the tumour or changes in corticosteroid dose. Failure to return for evaluation as a result of death or deteriorating condition. |

<sup>\*</sup> Increase in corticosteroid alone will not be taken into account in determining PD, in the absence of persistent clinical deterioration

NOTE: Patients with non-measurable disease only cannot have a complete response, the best

#### Response Assessment for Neuroblastoma

response possible is stable disease.

Protocol: ACCT008/ASSG35

The revised International Neuroblastoma Response Criteria (INRC) will be used to evaluate tumour response. Overall response will be defined by the response of the individual components – soft tissue, bone, and bone marrow disease per the investigator at each imaging timepoint..

| Overall Response | Criterion |
|---|---|
| Complete Response (CR) | All components meet criteria for CR |
| Partial Response (PR) | PR in at least one component and all other components are either CR, MD (minimal disease, bone marrow), PR (soft tissue or bone), or not involved* (NI); no component with PD |
| Minor Response (MR) | PR or CR in at least one component but at least one other component with SD; no component with PD SD in one component with no better than SD or not |
| Stable Disease (SD) | involved* (NI) in any other component; no component with PD |
| Progressive Disease (PD) | Any component with PD |

<sup>\*</sup> Site not involved at study entry and remains uninvolved.

See Appendix VI in protocol for more detail of Tumour Response Assessment Criteria and definitions.

#### 6.1 MAIN ANALYSIS

#### 6.1.1 Clinical Benefit rate

#### **Estimand**

**Population**: All patients eligible and enrolled into trial with MRT/ATRT (strata 1), osteosarcoma (strata 2), or neuroblastoma (strata 3).

**Treatment**: Panobinostat, dosing as per protocol.

Outcome: Efficacy as measured by Clinical Benefit Rate (CBR)

**Summary measure**: Clinical benefit rate (CBR) is the proportion of patients with an overall response of stable disease or better at MRI/CT imaging at 6- and 12-months post treatment commencement. CBR proportion (95% CI) and number will be reported for each disease strata.

Stable disease is defined as MRT/ATRT/Osteosarcoma with CR/PR/MR/SD/ overall response. Neuroblastoma with CR/PR/SD or Non-CR/Non-PD overall response.

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

6- and 12- months post treatment commencement will be the overall response disease assessment closest to 6 or 12 months ( $30.437 \, days \times (6 \, or \, 12) = XX \, days$ ) after the patient first dose (day 1 course 1) or enrolled date if patient didn't start treatment.

### **Intercurrent Events**

#### **Potential intercurrent events:**

Patient comes off study or treatment due to toxicity before an event is observed. Patient comes off study or treatment to receive another treatment.

## Strategy for handling intercurrent event:

**Treatment policy** 

CBR will be estimated for patients regardless early treatment or trial termination..

## **Sensitivity Analysis**

**Composite Strategy** 

Composite strategy includes early treatment termination as no benefit (not stable disease).

#### **Calculation of Estimand**

The CBR and 95%CI will be estimated using Statas ci proportions command.

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

## 7. EXPLORATORY OUTCOMES

## 7.1 COMPARISON TO HISTORICAL DATA

Comparison of NORTH ATRT patients to historical control will be outlined in a separate document. This will be attached as an appendix to this SAP once complete.

## 8. MISSING DATA

The number of patients with missing disease response/imaging at each timepoint will be listed by disease strata and any reasons provided listed.

Last patient contact and timepoint censored will be summarised and listed for patients.

## 9. LISTINGS, TABLES AND FIGURES

# 9.1. LIST OF LISTINGS

| Listing 1 | Listing of patient and disease characteristics at baseline |
|-----------|------------------------------------------------------------|
| Listing 2 | Listing of protocol deviations by strata |
| Listing 3 | Concomitant Medication |

## 9.2. LIST OF TABLES

| Table 1 | Patient recruitment and screening |
|----------|------------------------------------------------------------|
| Table 2 | Disease Characteristics at Baseline |
| Table 3 | Patient Characteristics at Baseline |
| Table 4 | Summary of treatment courses and follow up completed. |
| Table 5 | Number of patients completed each course by disease strata |
| Table 6 | Panobinostat Dosing by disease strata |
| Table 7 | Panobinostat Compliance by disease strata |
| Table 8 | Primary Outcome: Event free Survival |
| Table 9 | Primary Outcome: Overall Survival |
| Table 10 | Adverse Event Summary |
| Table 11 | Dose Limiting Toxicities |
| Table 12 | Secondary Outcome: Clinical Benefit Rate |
| Table 13 | Missing data |
| Table 14 | Censored Table |

# 9.3. LIST OF FIGURES

| Figure 1 | CONSORT diagram- NORTH trial |
|----------|------------------------------|
| Figure 2 | Kaplan-Meier curves of EFS |
| Figure 3 | Kaplan-Meier curves of OS |

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

#### **REFERENCES**

1. Simon R. Optimal Two Stage Designs for Phase II Clinical Trials. Controlled Clinical Trials. 1989; (10): 1-10.

- Food and Drug Administration. Center for Drug Evaluation and Research, Center for Biologics Evaluation and Research 2021. Guidance Document: E9(R1) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials. Guidance for Industry <a href="https://www.fda.gov/regulatory-information/search-fdaguidance-documents/e9r1-statistical-principles-clinical-trials-addendum-estimandsand-sensitivity-analysis-clinical">https://www.fda.gov/regulatory-information/search-fdaguidance-documents/e9r1-statistical-principles-clinical-trials-addendum-estimandsand-sensitivity-analysis-clinical</a>
- Food and Drug Administration. Oncology Center of Excellence. 2018. Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics Guidance for Industry. <a href="https://www.fda.gov/media/71195/download">https://www.fda.gov/media/71195/download</a>
- Food and Drug Administration. Center for Drug Evaluation and Research (CDER). 2015.
   Clinical Trial Endpoints for the Approval of Non-Small Cell Lung Cancer Drugs and
   Biologics Guidance for Industry. <a href="https://www.fda.gov/media/116860/download">https://www.fda.gov/media/116860/download</a>
- Pytynia KB, Grant JR, Etzel CJ, Roberts D, Wei Q, Sturgis EM. Matched Analysis of Survival in Patients With Squamous Cell Carcinoma of the Head and Neck Diagnosed Before and After 40 Years of Age. Arch Otolaryngol Head Neck Surg. 2004;130(7):869– 873. doi:10.1001/archotol.130.7.869
- 6. Rodríguez Germán. Cox Proportional Hazards with Two Groups. Survival Analysis. https://grodri.github.io/survival/cox

 Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan

## APPENDIX A. EXAMPLE TABLES AND FIGURES

**Listing 1:** Patient and disease characteristics at baseline



 Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

Table 1- Patient recruitment

Disease Type

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

| n | n | n |
|---|--------|---------|
| n | n | n |
| n | n | n |
| n | n | n |
| n | n | n |
| | n<br>n | n n n n |

recruitment prior to the initial efficacy analysis due to Panobinostat supply analysis due to Panobinostat supply

**Table 2** – Disease Characteristics at Baseline

| | | | Atypical Teratoid | | |
|---|---|---|---|---|---|
| | | Malignant Rhabdoid Tumor | Rhabdoid Tumor | | |
| Disease | MRT/ATRT | (MRT) | (ATRT) | Osteosarcoma | Neuroblastoma |

MRT/ ATRT

Neuroblastoma<sup>†</sup> Osteosarcoma<sup>†</sup>

| | n | n | n | n | n |
|---|---|---|---|---|---|
| Event | Newly Diagnosed n(%) | Newly Diagnosed n(%) | Newly Diagnosed n(%) | Un-resectable lesion n(%) | Refractory n(%) |
| | Relapsed n(%) | Relapsed n(%) | Relapsed n(%) | Relapsed n(%) | Relapsed n(%) |
| | | | | | , |
| Relapse no. | 1 n(%) | 1 n(%) | 1 n(%) | 1 n(%) | 1 n(%) |
| Kelapse IIO. | 2 n(%) | 2 n(%) | 2 n(%) | 2 n(%) | 2 n(%) |
| | 3 n(%) | 3 n(%) | 3 n(%) | 3 n(%) | 3 n(%) |
| Status | 4 n(%) | 4 n(%) | 4 n(%) | 4 n(%) | 4 n(%) |
| Status | | CR (n%) | CR (n%) | CR (n%) | CR (n%) |
| | CR (n%) | SD (%) | SD (%) | SD (%) | SD (%) |
| SI | 0 (%) | | | | |
| CNS involveme | ent n(%) | n(%) | n(%) | n(%) | n(%) |
| | CR n(%) | CR n(%) | CR n(%) | CR n(%) | CR n(%) |
| Best Respons | · · | SD n(%) | SD n(%) | SD n(%) | SD n(%) |
| · | PR n(%) | PR n(%) | PR n(%) | PR n(%)n(%) | PR n(%) |
| <b>Surgery</b> n( | %) n(%) n(%) | n(%) n(%) | | | |
| Chemothera | <b>py</b> n(%) | n(%) | n(%) | n(%) | n(%) |
| | RT n(%) | Brain or skull n(%) | Brain or skull n(%) | Brain or skull n(%) | Brain or skull n(% |
| | Spine n(%) | Spine n(%) | Spine n(%) | Spine n(%) | Spine n(%) |
| RT | Chest/thorax n(%) | Chest/thorax n(%) | Chest/thorax n(%) | Chest/thorax n(%) | Chest/thorax n(% |
| | Abdomen n(%) | Abdomen n(%) | Abdomen n(%) | Abdomen n(%) | Abdomen n(% |
| | Tibia n(%) | Tibia n(%) | Tibia n(%) | Tibia n(%) | Tibia n(%) |
| RT Total Dose (Gy) | mean(min-max) | mean(min-max) | mean(min-max) | mean(min-max) | mean(min-max |
| | BMT/PBSC n(%) | BMT/PBSC n(%) | BMT/PBSC n(%) | BMT/PBSC n(%) | BMT/PBSC n(% |
| Other treatment | | | | | |
| | Other (list) n(%) | Other (list) n(%) | Other (list) n(%) | Other (list) n(%) | Other (list) n(% |

**Table 3** – Patient Characteristics at Baseline

Protocol: ACCT008/ASSG35

| | | Malignant Rhabdoid | Atypical Teratoid<br>Rhabdoid Tumor | | |
|---|---|---|---|---|---|
| Disease | | | | | |
| MRT/ATRT | mean (min-max) | mean (min-max) | mean (min-max) | mean (min-max) | X,X |
| Tumor (MRT) | Male n(%) Female n(%) | Male n(%) Female n(%) | Male n(%) Female n(%) | Male n(%) Female n(%) | VV |
| (ATRT) | Male II(%) FeIIIale II(%) | Male 11(%) remaie 11(%) | iviale II(%) FeIIIale II(%) | Male II(%) FeIIIale II(%) | X,X |
| Osteosarcoma | | Asian n(%) Black n(%) | Asian n(%) Black n(%) | | |
| euroblastoma | Asian n(%) Black n(%) | Caucasian n(%) | Caucasian n(%) | Asian n(%) Black n(%) | |
| Age | Caucasian n(%) Unknown | Unknown n(%) Other | Unknown n(%) Other | Caucasian n(%) Unknown | X,X |
| Sex | n(%) Other n(%) | n(%) | n(%) | n(%) Other n(%) | |
| | Neit | Neither Aboriginal or<br>Torres Strait Islander<br>her Aboriginal or Neither A | Neither Aboriginal or<br>Torres Strait Islander<br>Aboriginal or n(%) | n(%) | |
| | | her Aboriginal or Neither A | Aboriginal or n(%) | · · | |
| | Torres Strait Islander n(%) | | | Torres Strait Islander n(%) | |
| | | Both Aboriginal or | Both Aboriginal or | | |
| | Both Aboriginal or Torres | | | Both Aboriginal or Torres | |
| | 6 (01) | Torres Strait Islander | Torres Strait Islander | | |
| | Strait Islander n(%) | Strait Islander n(%) | X,X n(%) n(%) | AL (0/) | |
| | Aboriginal n(%) | | 41 (0/) | Aboriginal n(%) | |
| | T Charle I-l (2/) | Aboriginal n(%) | Aboriginal n(%) | Tamas Studit Islandan (00) | |
| | Torres Strait Islander n(%) | Tamas Chusin Island | Tamas Charle Iala | Torres Strait Islander n(%) | |
| | 11 | Torres Strait Islander | Torres Strait Islander | | |
| | | , , | own n(%) n(%) n(%) | | |
| ın | digenous status Unknown n | (70) | Unknown n(%) | | |

mean (min-max)

mean (min-max)

X,X

mean (min-max)

Performance Score mean (min-max)

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

Listing 2: List of protocol deviations, by site.

| Site | Deviation | Timepoint | Date |
|------|-----------|-----------|------|
| x | x | x | x |

**Table 4** – Summary of treatment courses and follow up completed.

| | MRT/ATRT | Osteosarcoma | Neuroblastoma |
|---|---|---|---|
| Number of completed courses of treatment | mean(min-max) | mean(min-max) | X,X |
| Time in Follow Up (weeks) Mean and range (min-max) | mean(min-max) | mean(min-max) | X,X |

**Table 5** – Number of patients completed each course by disease strata.

| | | Number of | Number of Patients who completed Course (28 days) | | |
|---|---|---|---|---|---|
| | | | | Number of Early | <b>Early Termination</b> |
| MRT/ATRT | n | n | n | n | Х |
| Osteosarcoma | n | n | n | n | X |
| Neuroblastoma | n | n | n | n | X |
| Terminations | n | n | n | n | X |
| Reason | n | n | n | n | X |
| Course 1 | n | n | n | n | X |
| Course 2 | n | n | n | n | X |
| Course 3<br>Course 4 | n | n | n | n | X |
| Course 5 | n | n | n | n | X |
| Course 6 | n | n | n | n | X |
| Course 7 | n | n | n | n | X |
| Course 8 | n | n | n | n | X |
| Course 9 | | | | | |
| Course 10 | | | | | |
| Course 11 | | | | | |
| Course 12 | | | | | |

**Table 6** – Panobinostat Dosing by Course and Disease strata

## Patient Dosing (mg/m2)

| _ | MRT/ATRT | Osteosarcoma | Neuroblastoma |
|--------------|--------------|--------------|---------------|
| Course 1 | mean(minmax) | mean(minmax) | X,X |
| Course 2 | mean(minmax) | mean(minmax) | X,X |
| Course 3 | mean(minmax) | mean(minmax) | X,X |
| Course 4 | mean(minmax) | mean(minmax) | X,X |
| Course 5 | mean(minmax) | mean(minmax) | X,X |
| Course 6 | mean(minmax) | mean(minmax) | X,X |
| Course 7 | mean(minmax) | mean(minmax) | X,X |
| Course 8 | mean(minmax) | mean(minmax) | X,X |
| Course 9 | mean(minmax) | mean(minmax) | V V |
| Course<br>10 | | | X,X |
| Course | mean(minmax) | mean(minmax) | X,X |
| 11<br>Course | mean(minmax) | mean(minmax) | X,X |
| 12 | mean(minmax) | mean(minmax) | X,X |
| Гable 7 — | | | |

Course and Disease strata

| | Dose (mg/m2) | Days Compliant | Total Days |
|--------------|---------------|----------------|---------------|
| MRT/ATRT | mean(min-max) | mean(min-max) | mean(min-max) |
| Osteosarcoma | mean(min-max) | mean(min-max) | mean(min-max) |
| | <i>X, X</i> | X, X) | X, X) |

## Neuroblastoma

Mean and range (min-max)

**Listing 3:** Concomitant Medication

Sorted by disease strata.

| Disease Strata | <b>Medication Name</b> | <b>Medication Reason</b> |
|----------------|------------------------|--------------------------|
| MRT/ATRT | X | Х |

| Protocol: ACCT008/ASS | G35 NORTH: Stat | istical Analysis Plan |
|---|---|---|
|---|---|---|

| MRT/ATRT | x | X |
|---------------|---|---|
| MRT/ATRT | x | X |
| Osteosarcoma | x | X |
| Osteosarcoma | x | X |
| Osteosarcoma | x | X |
| Neuroblastoma | x | X |
| Neuroblastoma | x | X |
| Neuroblastoma | x | X |
| | l | |

**Table 8** - Primary Endpoint: Event Free Survival

## **Primary Outcome- EFS**

| x(95%CI) | x(95%CI) | Х |
|-------------------------------------|------------|----|
| x(min-max) | x(min-max) | NA |
| x(95%CI) | x(95%CI) | X |
| x(min-max) | x(min-max) | NA |
| Proportion<br>(95%CI) | | |
| Proportion(95%CI) Proportion(95%CI) | | |
| 11000111011(33/001) | | |

MRT/ATRT Osteosarcoma Neuroblastoma

Overall EFS (95%CI)

Median EFS, months (95%CI)

**Sensitivity Analysis - Composite Strategy** 

Overall EFS (95%CI)

Median EFS, months (95%CI)

## **Subgroup Analysis**

Age at enrolment (<36 months vs. (≥36 months)

Radiation therapy (RT vs. no RT)

Up to 2 years post study enrolment

Table 9: Primary Endpoint: Overall Survival

#### Disease status

Overall Survival (95%CI)
Median overall survival, months (95%CI)
Number of deaths

## **Subgroup Analysis**

Age at enrolment (<36 months vs. (≥36 months)
Radiation therapy (RT vs. no RT)
Disease Status

Up to 2 years post study enrolment

| Ī | x(95%CI) | x(95%CI) | |
|---|---|---|---|
| | x(95%CI) | x(95%CI) | |
| | n<br>Proportion<br>(95%CI)<br>Proportion<br>(95%CI)<br>Proportion<br>(95%CI) | n | n |
| ı | (33/00/) | | |

## **Table 10** - Treatment-Related Adverse Events

Treatment-Related Adverse Events
Toxicity (CTCAE Any Grade v4.0)

| _ | | | | | |
|---------|------|---|---|---|---|
| | n(%) | n | n | n | n |
| Grade 4 | n(%) | n | n | n | n |
| event | n(%) | n | n | n | n |
| event | | | | | |
| event | n(%) | n | n | n | n |
| event | | | | | |

Event Grade 1 Grade 2 Grade 3

**Table 11** – Dose Limiting Toxicities

**Dose Limiting Toxicity Adverse Events** 

Toxicity (CTCAE v4.0)

1 n
2 n
3 n
4 n
Grade Frequency

event event event

Table 12- Secondary Outcome: Clinical Benefit Rate

## **Secondary Outcome- Clinical Benefit Rate**

| x(95%CI) x(95%CI) x(95%CI) x(95%CI) x(95%CI) x x(95%CI) x | na |
|---|---|
| x(95%CI) x(95%CI) x | |
| x(95%CI) x(95%CI) x | |

Protocol: ACCT008/ASSG35 NORTH: Statistical Analysis Plan 

CBR at 6 months %(95%CI)
CBR at 12 months %(95%CI)
Sensitivity Analysis - Composite Strategy
CBR at 6 months %(95%CI)
CBR at 12 months %(95%CI)

Table 13 - Missing Data

## Missing Outcome Data

| Disease Strata | Data Missing | Reason missing |
|----------------|------------------------|------------------------|
| MRT/ATRT | Disease Assessment | Scan not performed (n) |
| Osteosarcom | a Lesions not measured | on scan (n) |
| Neuroblastoma | | Other reasons (n) |

Table 14 -Censored table

| Study ID | Last patient contact (Timepoint) | Censored (Y/N) |
|----------|----------------------------------|----------------|
| 1 | Week 6 | Y |
| 2 | Follow-up | N |

# STATISTICAL REPORT

Final Audit Report 2025-01-06

Created: 2025-01-06

By: Alannah Rudkin (alannahrudkin@gmail.com)

Status: Signed

Transaction ID: CBJCHBCAABAAW\_WVYuYZRonABUXmlJo-ObbJ8Z7yT7TD

# "STATISTICAL REPORT" History

Document created by Alannah Rudkin (alannahrudkin@gmail.com) 2025-01-06 - 5:02:51 AM GMT- IP address: 165.225.226.227

- Document emailed to A/Prof Jayesh Desai (jayesh.desai@petermac.org) for signature 2025-01-06
  - 5:02:57 AM GMT
- Email viewed by A/Prof Jayesh Desai (jayesh.desai@petermac.org) 2025-01-06 5:07:30 AM GMT- IP address: 121.221.169.186
- Document e-signed by A/Prof Jayesh Desai (jayesh.desai@petermac.org)

  Signature Date: 2025-01-06 5:48:15 AM GMT Time Source: server- IP address: 203.4.166.50
- Agreement completed.

